CLINICAL TRIAL: NCT02766101
Title: Can a Physical Activity Program Implemented at a Therapeutic School Promote Emotional Regulation and School Success in Socially and Emotionally Vulnerable Children?
Brief Title: Manville Moves: an Exercise Intervention for Behavioral Regulation Among Children With Behavioral Health Challenges
Acronym: MM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Judge Baker Children's Center (Other)
Responsible Party: Principal Investigator, Kirsten Davison, Associate Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-2312
Record Dates: First submitted 2016-04-25; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Autistic Disorder; Attention Deficit and Disruptive Behavior Disorders; Anxiety Disorders; Mood Disorders; Conduct Disorder; Oppositional Defiant Disorder
MeSH Terms: conditions — Autistic Disorder; Attention Deficit and Disruptive Behavior Disorders; Anxiety Disorders; Mood Disorders; Conduct Disorder; Oppositional Defiant Disorder

ARMS (2):
- Aerobic Exergaming PE (Experimental): Progressive aerobic curriculum utilizing virtual reality exergaming stationary bicycles. Classes held 2 times per week for 30-40 minutes, aerobic exercise beginning at 10 minutes at moderate to vigorous intensity and building to 20 minutes plus.
  Interventions: Behavioral: Aerobic Exergaming PE Curriculum
- Standard PE (Active Comparator): Traditional PE focused on gross motor skill and sports skill acquisition, and team building. Typically non-aerobic.
  Interventions: Behavioral: Standard PE

INTERVENTIONS:
Behavioral: Aerobic Exergaming PE Curriculum — Sustained aerobic exercise.
  Arms: Aerobic Exergaming PE
Behavioral: Standard PE — Non-aerobic skill building.
  Arms: Standard PE

SUMMARY:
The purpose of this study is to examine whether an exergaming, aerobic physical education (PE) curriculum is acceptable and elicits improvements in behavioral self-regulation and classroom functioning among children with behavioral health challenges attending a therapeutic day school. After following an approved consent/assent process, children attending the school were randomized by classroom to take part in either 7 weeks of the experimental PE curriculum, or 7 weeks of the standard PE curriculum; after a 10 week washout period, children then crossed over into the other arm.

ELIGIBILITY:
Inclusion Criteria:

* Attending the Manville School at the time of study initiation

Exclusion Criteria:

* Medical exemption from physical education classes
* Parental opt out from physical education classes

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in Minutes and Number of Disciplinary Time Out of Class Events (classroom functioning) | Assessed Daily for 14 weeks (7 weeks in intervention arm and 7 weeks in control arm)
  Recording of student number of times and total minutes per day asked to leave the classroom due to disruptive or aggressive behavior. This outcome measure is recorded at the time of event on a mobile survey platform by the present classroom counselor. The measure may be dichotomized into clinical thresholds of time out of class either disruptive or preclusive of learning. A common measurement of classroom functioning in therapeutic school environments.
Change in Conners Abbreviated Teacher Rating Scale score (behavioral dysregulation: impulsivity/emotional lability) | Assessed Daily for 14 weeks (7 weeks in intervention arm and 7 weeks in control arm)
  Recording of classroom counselor assessment of student impulsivity/hyperactivity and emotional lability using the Conners Abbreviated Teacher Rating Scale 10-item (CATRS-10). CATRS-10 is a commonly used and validated screening instrument for behavioral problems related to inattention, impulsivity/hyperactivity and emotional lability. Classroom counselors completed the CATRS-10 at the end of each school day for each student. The instrument consists of 10 statements regarding the child's behavior rated on a 4-point Likert scale, with a possible total score from 0 to 30. A score of 15 or higher has been the standard for screening children with symptomology at a level of clinical concern.Equivalent screening thresholds were used for the emotional lability subscale (≥6 out of possible 12) and impulsivity subscale (≥9 out of possible 18). Thus this outcome measure can also be dichotomized for analytical and clinical interpretation purposes.

CONTACTS AND LOCATIONS:
Locations (1):
- Judge Baker Children's Center, Manville School, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Davison K, Bowling A, Garcia J, Wood B, Hermesch R, Prince J, Hayes A, Kow R, Newlan S, Slavet J. A cybercycling intervention to improve behavioral regulation and classroom functioning among children with behavioral health disorders: Pragmatic randomized trial design for Manville Moves. Contemp Clin Trials. 2016 Jul;49:40-6. doi: 10.1016/j.cct.2016.05.008. Epub 2016 May 31. PMID 27261171